CLINICAL TRIAL: NCT01197664
Title: A Pilot Study of Paricalcitol Synergism in Conjunction With Standard-of-Care Chemo-Radiation for Resectable Rectal Cancers
Brief Title: Paricalcitol, Fluorouracil, and Radiation Therapy in Treating Patients With Rectal Cancer That Can Be Removed in Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to funding issues
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00013006; NCI-2011-02409 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 54110 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Mucinous Adenocarcinoma of the Rectum; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIB Rectal Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — paricalcitol; Radiotherapy; Radiation; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (paricalcitol and chemoradiotherapy) (Experimental): Patients receive paricalcitol PO daily. Patients also receive standard care chemoradiotherapy with fluorouracil PO.
  Interventions: Drug: paricalcitol; Radiation: radiation therapy; Other: laboratory biomarker analysis; Drug: fluorouracil
- Arm II (chemoradiotherapy) (Active Comparator): Patients receive standard care chemoradiotherapy as in Arm I.
  Interventions: Radiation: radiation therapy; Other: laboratory biomarker analysis; Drug: fluorouracil

INTERVENTIONS:
Drug: paricalcitol — Given PO
  Other Names: Zemplar
  Arms: Arm I (paricalcitol and chemoradiotherapy)
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies
Drug: fluorouracil — Given PO
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
This randomized pilot clinical trial studies the side effects of giving paricalcitol together with fluorouracil and radiation therapy in treating patients with rectal cancer that can be removed in surgery. Paricalcitol may help rectal cancer cells become more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x rays to kill tumor cells. It not yet known if chemotherapy and radiation therapy are more effective with or without paricalcitol in treating rectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate toxicity and tolerability of oral paricalcitol at 2 μg/day when co-administered with oral 5-fluorouracil (fluorouracil)-based chemoradiation in patients with histologically confirmed, resectable T3-T4 adenocarcinoma of rectal mucosal origin or node-positive disease with no known distant metastases.

SECONDARY OBJECTIVES:

I. To study the biologic effects of oral paricalcitol in addition to oral 5-fluorouracil chemoradiation on Vitamin D receptor staining, MIB-1, Caspase 3, P 21, and Bax protein expression in these patients.

II. To identify patterns of gene expression in tumor samples of patients who receive chemo radiation with and without Paricalcitol supplementation using gene microarray technology.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paricalcitol orally (PO) daily. Patients also receive standard care chemoradiotherapy with fluorouracil PO.

ARM II: Patients receive standard care chemoradiotherapy as in Arm I.

In both arms, treatment continues until surgical resection in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histologically confirmed T3-T4 adenocarcinoma of rectal mucosal origin or node positive, with no confirmed distant metastases, and that has been shown to be resectable Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Leukocytes >= 3,000/mcL Absolute neutrophil count >= 1,500/mcL Platelets >= 100,000/mcL Total bilirubin within normal institutional limits Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal Patients must not have deficient levels of Vitamin D, 1, 25 Hydroxy as defined by the institution (this allows patients with normal vitamin D or insufficient vitamin D) Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

No prior pelvic radiation therapy or chemo-radiation to the rectum; no chemo-radiation for any other reason in the last 8 weeks Patients may not be receiving any other investigational agents Patients with a history of or current hypercalcemia may not be enrolled in this study History of allergic reactions attributed to compounds of similar chemical or biologic composition to paricalcitol Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements Pregnant women and nursing mothers are excluded from this study because the adverse effects on the fetus from chemo radiation Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with these agents; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Toxicity and tolerability of the paricalcitol regimen, as measured by calcium levels | Assessed up to surgical resection
  Calcium levels will be noted on a weekly basis during chemoradiotherapy and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

SECONDARY OUTCOMES:
Biologic effects of oral paricalcitol with oral fluorouracil chemoradiation on vitamin D receptor staining, MIB-1, caspase 3, p 21, and bax protein expression | Baseline
Biologic effects of oral paricalcitol with oral fluorouracil chemoradiation on vitamin D receptor staining, MIB-1, caspase 3, p 21, and bax protein expression | Day 14
Biologic effects of oral paricalcitol with oral fluorouracil chemoradiation on vitamin D receptor staining, MIB-1, caspase 3, p 21, and bax protein expression | At surgical resection
Patterns of gene expression in tumor samples of patients who receive chemoradiation with and without paricalcitol | Baseline
Patterns of gene expression in tumor samples of patients who receive chemoradiation with and without paricalcitol | Day 14
Patterns of gene expression in tumor samples of patients who receive chemoradiation with and without paricalcitol | At surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: George Yacoub, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States